CLINICAL TRIAL: NCT06055218
Title: Evaluation of the Performance of Novel Molecular Point of Care Diagnostics for SARS-CoV-2
Brief Title: COVID-19 Novel Molecular Point of Care Diagnostics Evaluation
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CV010
Record Dates: First submitted 2023-09-25; First posted 2023-09-26 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Point estimates of sensitivity and specificity of molecular POC platforms for SARS-CoV-2, with 95% confidence intervals, using RT-PCR as reference standard.

DETAILED DESCRIPTION:
The aim of this study is to independently evaluate the performance of novel molecular point-of-care (POC) assays for the direct detection of SARS-CoV-2 nucleic acid (RNA) in comparison to the current reference standard, laboratory-based real-time reverse-transcription PCR (RT-PCR), for use to diagnose COVID-19, a serious and sometimes fatal respiratory infection caused by the coronavirus SARS-CoV-2. A total of 3 molecular POC devices, detecting SARS-CoV-2 and other viral pathogens, have been selected by FIND through open calls for expressions of interest. These are Covid/RSV/Flu Nudge Test (DnaNudge Ltd, Nudge test from hereon), Test Kit for SARS-CoV-2 RNA Detection in Biological Material Using PCR Method (Mirai Genomics, Mirai test from hereon) and GenomEra (Abacus Diagnostica Oy, GenomEra test from hereon). Other molecular POC devices currently in the late development stage may become available for assessment of clinical performance at later time, should these pass FIND's selection criteria.

The COVID-19 pandemic has rapidly spread across the globe. As of 3 October 2022, there are approximately a total of 623 million confirmed cases reported worldwide, that resulted in a total of 6.55 million deaths. The current weekly incidence is on average 1 million new cases. However, the consensus among public health officials is that the number of infected individuals is far higher. Given the wide range of possible symptoms and the potential for transmission before individuals are aware that they are infected, exposure to SARS-CoV-2 is a particular hazard for health care providers. Though diagnostic capacity has greatly improved due to the introduction of novel antigen rapid diagnostic tests (Ag RDT), long turnaround times for results of the current reference standard for testing (RT-PCR) is still a major challenge. This impacts on the ability of public health officials to track and contain the disease. The lack of capacity, in turn, is due in part to the logistic challenges and global reagent shortages faced by laboratories attempting to implement new RT-PCR assays for SARS-CoV-2.

Rapid sample-in-answer-out molecular POC devices, if shown to have sufficient accuracy to aid in clinical decision-making, could contribute substantially to control the disease spread globally. Molecular POC devices might provide a source of immediate diagnostic testing in low-and middle-income countries unable to implement RT-PCR due to lack of sample transport and storage facilities at local laboratories.

ELIGIBILITY:
Inclusion Criteria: Participants and specimens are eligible to be included in the study only if all the following inclusion criteria apply:

* Adult individuals (≥18 years of age) with symptoms suggesting plausible COVID-19 infection (as per WHO or national clinical case definitions)
* Individuals who have voluntarily given written consent to participate in this study or who have given their written consent for their specimen to be used for future research studies
* Individuals able to provide the specimens required for the study

Exclusion Criteria:

* Individuals on oxygen therapy
* Individuals with recent history of excessive nose bleeds
* Individuals with hemodynamic instability as determined by their treating physician
* Individuals already enrolled in other clinical studies, where similar respiratory specimens are collected on the same day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specimens to be tested for this study must originate from adult symptomatic individuals (≥ 18 years old) suspected to have COVID-19 (as per national or WHO case definitions).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specitivity | at enrollement
  Point estimates of sensitivity and specificity of molecular POC platforms

SECONDARY OUTCOMES:
Sensitivity and specificity in specific subgroups | at enrolment
  Point estimates of sensitivity and specificity of molecular POC platforms for SARS-CoV-2, with 95% confidence intervals, using RT-PCR as reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Escadafal, Study Chair — FIND Diagnostics
Locations (3):
- University Hospital of Geneva, Geneva, Switzerland
- Central Public Health Laboratories, Kampala, Uganda
- Liverpool school of Topical Medicine, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No